CLINICAL TRIAL: NCT00554957
Title: Perception of Musculoskeletal Injury in Professional Dancers, an International Comparison
Brief Title: Perception of Musculoskeletal Injury in Professional Dancers
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Southern Denmark (Other); Lund University (Other); Hadassah Medical Organization (Other)
Responsible Party: Craig Jacobs, Artists' Health Centre Foundation Research Programme
Other Study IDs: 06-0930-AE
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Musculoskeletal System; Disability Evaluation; Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- NBC: All dancers with the National Ballet of Canada will be given the opportunity to participate in the study.
- TDT: All dancers with the Toronto Dance Theatre will be given the opportunity to participate.
- KDC: All members of the Kibbutz Contemporary Dance company will be given the opportunity to participate.
- BDC: All dancers with the Batsheva Dance Company or Ensemble will be given the opportunity to participate.
- RSB: All dancers with the Royal Swedish Ballet will be given the opportunity to participate.
- RDB: All dancers with the Royal Danish Ballet will be given the opportunity to participate.

SUMMARY:
The annual frequency of injury among dancers has been reported to range between 23-84% while as many as 95% of professional dancers have ongoing pain. The discrepancy between the number of reported injuries and the amount of pain reported at any given time could be related to the definition of injury, or how dancers' themselves perceive injury with respect to pain and activity limitation thresholds. For many reasons, dancers may be dancing through or past what health care providers may conceive as injury. This can put them at risk of further or chronic injury. The purpose of this study is to understand at which point pain limits a dancer's ability to continue to perform and whether this is influenced by available medical services, a supportive dance environment, or other factors. In addition, the issue of non-reporting of injuries will be studied. This is very important as this will affect all measures of injury frequency and risk for dancers.

DETAILED DESCRIPTION:
Brief Rationale and Objective:

The annual frequency of injury among dancers has been reported to range between 23-84% while as many as 95% of professional dancers have ongoing pain. The discrepancy between the number of reported injuries and the amount of pain reported at any given time could be related to the definition of injury, or how dancers' themselves perceive injury with respect to pain and activity limitation thresholds. For many reasons, dancers may be dancing through or past what health care providers may conceive as injury. This can put them at risk of future recurrent or chronic injury. The purpose of this study is to gain insight into professional dancers' perception of musculoskeletal (MSK) injury in order to understand at which point pain limits a dancer's ability to continue to perform and to determine what factors influence a dancer's perception of injury and decision to seek or not seek care. We will investigate whether this is influenced by available medical services, a supportive dance environment, or other factors. In addition, the issue of non-reporting of injuries will be studied. This is very important because it affects all measures of injury frequency and risk for dancers.

Research Questions:

The purpose of this study will be to answer the following questions: 1) What is the prevalence of MSK injury-related pain in the dance company? 2) What are the pain and activity limitation thresholds for a dancer to consider him/herself injured? 3) What factors are associated with considering him/herself injured? 4) What constitutes a major or a minor injury to a dancer? 5) How are dancers reporting their injuries? 6) How many dancers are not reporting their injuries and what are the reasons? 7) Do the answers to the above questions differ between countries (Canada, Israel, Sweden, Denmark) that have varying levels of social and medical support for dancers?

Design and Methodology:

Design: Cross-sectional survey. Study Population: All dancers employed by: The National Ballet of Canada, Toronto Dance Theatre, Batsheva Dance Company and Ensemble (Israel), The Kibbutz Contemporary Dance Company (Israel), the Royal Swedish Ballet (Sweden), and the Royal Danish Ballet (Denmark). Total approximate number of participants is 294. Methods: Two questionnaires will be distributed to participants. The Self-Estimated Functional Inability because of Pain (SEFIP) questionnaire is a validated tool for dancers which has shown good agreement with actual pain found on physical examination. The SEFIP will be used in order to measure pain and functional deficits. An additional questionnaire will be used to gain further information regarding the above research questions. There will be an area for the dancers to include any additional comments in relation to these subjects in order to capture further qualitative data. Data Analysis: Descriptive statistics will be reported in the form of percentages and means with standard deviations. Non-parametric tests will be used to analyze categorical variables. 95% confidence intervals will be reported for each analysis. The qualitative data captured in the open-ended questions will be analyzed for common themes in order to provide further explanation for the quantitative data as well as to provide additional information for further research.

Significance:

A recent systematic review of the dance injury literature stressed the necessity of a standardized definition of injury for future research studies involving dancers. This study will attempt to address the dancer's perspective in regards to perception of injury. We believe this international study will provide insight into the frequency and reporting of dance-related pain and some potential factors that influence this. Ultimately, we hope to improve the health-related quality of life for dancers with musculoskeletal injury.

ELIGIBILITY:
Inclusion Criteria:

* All dancers employed by the National Ballet of Canada, Toronto Dance Theatre, Batsheva Dance Company and Ensemble, Kibbutz Contemporary Dance Company, the Royal Swedish Ballet, and the Royal Danish Ballet will be included in the study. Additional dance companies from Sweden, Israel, Denmark and Canada (and other countries) may be invited to participate. If so, then identical protocols will be followed for all companies.

Exclusion Criteria:

* Any dancer less than 18 years of age will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Professional Dancers
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2007-04; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Self Estimated Functional Inability because of Pain (SEFIP) Perception of Injury Questionnaire | Point prevalence

SECONDARY OUTCOMES:
Numeric Rating Scale, Perception of Injury Questionnaire | Point prevalence

CONTACTS AND LOCATIONS:
Overall Officials: J. David Cassidy, PhD, DrMedSc, Principal Investigator — Toronto Western Research Institute; Craig L Jacobs, BFA, DC, Study Director — Toronto Western Research Institute
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Ramel EM, et al, Validation of a pain questionnaire (SEFIP) for dancers with a specially created test battery, Medical Problems of Performing Artists; December 1999.
- [Background] Tajet-Foxell B, Rose FD. Pain and pain tolerance in professional ballet dancers. Br J Sports Med. 1995 Mar;29(1):31-4. doi: 10.1136/bjsm.29.1.31. PMID 7788215
- [Background] Hamilton LH et al, Factors contributing to the attrition rate in elite ballet students, Journal of Dance Medicine and Science;1997;1(4).
- [Background] McNeal AP et al, Lower extremity alignment and injury in young, preprofessional college and professional ballet dancers, Part II: Dancer-reported injuries; Medical Problems of Performing Artists; June 1990.
- [Background] Ramel E, Moritz U. Self-reported musculoskeletal pain and discomfort in professional ballet dancers in Sweden. Scand J Rehabil Med. 1994 Mar;26(1):11-6. PMID 8023078
- [Background] Ramel E, Thorsson O, Wollmer P. Fitness training and its effect on musculoskeletal pain in professional ballet dancers. Scand J Med Sci Sports. 1997 Oct;7(5):293-8. doi: 10.1111/j.1600-0838.1997.tb00156.x. PMID 9338948